CLINICAL TRIAL: NCT01397188
Title: Effect of Monitoring of Pulse Index Continuous Cardiac Output on Shock Patients in ICU
Brief Title: Effect of Monitoring of Pulse Index Continuous Cardiac Output (PiCCO) on Shock Patients in Intensive Care Unit
Acronym: PiCCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li danyang (Other)
Responsible Party: Sponsor-Investigator, Li danyang, Dr, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19741016
Record Dates: First submitted 2011-07-08; First posted 2011-07-19 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Shock
Keywords: PiCCO
MeSH Terms: conditions — Shock | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PiCCO group (Experimental): Intervention: Device: Picco- thermodilution catheter
  Interventions: Device: PiCCO
- sham group (Sham Comparator): No PiCCO Intervention
  Interventions: Other: sham, no intervention

INTERVENTIONS:
Device: PiCCO — transpulmonary thermodilution technique
  Arms: PiCCO group
Other: sham, no intervention — no intervention
  Arms: sham group

SUMMARY:
PiCCO has become a widely used haemodynamic monitoring device in the management of shock patients in ICU patients nowadays. But the effects on outcome of use of Picco, such as hospital mortality, vasoactive agents-free days, intensive care unit, and mechanical ventilation-free days and change of lactate and BNP in shock patients has not been determined. Patients will be randomly assigned to a Picco group or the control group, hospital mortality, vasoactive agents-free days, intensive care unit, and mechanical ventilation-free days and change of lactate and BNP will be observed. The conclusion will supply evidence for the clinical effectiveness of Picco in shock patients.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients with shock: Mean arterial pressure (MAP) < 65 mmHg (< 8,7 kPa) or systolic arterial pressure (SAP) < 90 mmHg (< 12 kPa) or the need for vasopressor (Norepinephrine <0.05µg/kg/min) to support the MAP ≥ 65 mmHg (≥ 8,7 kPa) or the SAP ≥ 90 mmHg ≥ 12 kPa), when one of these criteria has lasted for 4 hours or longer

Exclusion Criteria:

* Age < 18 years
* Age > 85 years
* Pregnancy (positive pregnancy test in women of child bearing age)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
mortality at 28 days | 28 days
  mortality at 28 days after diagnosis of shock

SECONDARY OUTCOMES:
vasoactive agents-free days | 28 days
  vasoactive agents-free days: the number of days from day 1 to day 28 without use of vasoactive agents.
intensive care unit-free days | 28 days
  intensive care unit(ICU) free days, defined as the number of days from day 1 to day 28 without ICU stay.
mechanical ventilation-free days | 28 days
  ventilator free days: the number of days from day 1 to day 28 during which the patient breathed spontaneously
the change of lactate at 1,3,7 days after the insertion of the Picco catheter | 7 days
  blood samples will be taken before the insertion of the Picco catheter and everyday after the insertion, the change of lactate at 1,3,7 days after the insertion of the Picco catheter will be collected.
the change of B-Type Natruetic Peptide(BNP) at 1,3,7 days after the insertion of the Picco catheter | 7 days
  blood samples will be taken before the insertion of the Picco catheter and everyday after the insertion, the change of BNP at 1,3,7 days after the insertion of the Picco catheter will be collected.
mortality at 90 days | 90 days
  mortality at 90 days after diagnosis of shock

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital Medical College, Zhejiang University, Hangzhou, Zhejiang, China